CLINICAL TRIAL: NCT00499005
Title: Carbetocin Versus Syntometrine for the Third Stage of Labour Following Vaginal Delivery - A Double-blind Randomised Trial
Brief Title: Carbetocin Versus Syntometrine for the Third Stage of Labour
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Healthcare Group, Singapore (Other Government)
Responsible Party: Chong Yap Seng, MBBS, National HealthCare Group, Singapore
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: DSRB Ref: D/04/209; NHG-SIG/07059
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Postpartum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primi (Active Comparator)
  Interventions: Drug: Syntommetrine and Carbetocin
- Multi (Active Comparator)
  Interventions: Drug: Syntommetrine and Carbetocin

INTERVENTIONS:
Drug: Syntommetrine and Carbetocin — Syntommetrine 1ml and Carbetocin 100microgram
Drug: Syntommetrine and Carbetocin — Syntommetrine 1ml and Carbetocin 100micgrams

SUMMARY:
Intramuscular carbetocin is as effective as intramuscular syntometrine for the prevention of postpartum haemorrhage

DETAILED DESCRIPTION:
Postpartum haemorrhage(PPH)or excessive bleeding at or after childbirth is a potentially life threatening complication and is one of the major contributors to maternal mortality and morbidity worldwide (Lewis 2001).Among the various agents that have been studied in addition to the routine oxytocin and syntometrine (which has adverse effects),oxytocin agonist (carbetocin) appears to be the most promising for this indication(Chong 2004).

Carbetocin is a licensed medication for the use of prevention of postpartum haemorrhage in Singapore and many other countries. It is a long-acting synthetic octapeptide analogue of oxytocin with agonist properties.The clinical and pharmacological properties of carbetocin are similar to those of naturally occurring oxytocin. Like oxytocin, carbetocin binds to oxytocin receptors present on the smooth musculature of the uterus, resulting in rhythmic contractions of the uterus, increased frequency of existing contractions, and increased uterine tone. In pharmacokinetic studies, intravenous injections of carbetocin produced tetanic uterine contractions within two minutes, lasting six minutes, followed by rhythmic contractions for a further hour.Intramuscular injection produced tetanic contractions in less than two minutes, lasting about 11 minutes, and followed by rhythmic contractions for an additional two hours. The prolonged duration of activity after intramuscular compared with the intravenous carbetocin was significant(Hunter 1992). In comparison to oxytocin, carbetocin induces a prolonged uterine response when administered postpartum, in terms of both amplitude and frequency of contractions.

The potential advantage of intramuscular carbetocin over intramuscular oxytocin is its longer duration of action. Its relative lack of gastrointestinal and cardiovascular side-effects should also prove advantageous compared to syntometrine and other ergot alkaloids.

ELIGIBILITY:
Inclusion Criteria:

1. Any pregnant woman expected to deliver vaginally
2. Age more than 21 if not married
3. Ability to provide informed consent

Exclusion Criteria:

1. Multiple pregnancy
2. Patients with other risk factors for postpartum haemorrhage
3. Patients planning to have an elective caesarean section
4. History of vascular disease such as coronary artery disease
5. History of hypertension requiring treatment within the last 2 years
6. History of hepatic or renal disease
7. Known or suspected coagulopathy
8. History of hypersensitivity to oxytocin or carbetocin
9. Any condition where the use of syntometrine/carbetocin is contraindicated

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 720 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
1. Postpartum haemorrhage (less than or equal to 500 ml) 2. Postpartum haemorrhage (less than or equal to 1000ml) 3. Use of additional uterotonic therapy | Within 2 hours after delivery

SECONDARY OUTCOMES:
1. Adverse effects with the intervention which include headache, nausea, vomiting, elevation of blood pressure and retained placenta 2. Cost effectiveness analysis of the intervention | Within 2 hours after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Su Lin Lin, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore